CLINICAL TRIAL: NCT00308217
Title: The Examination of Outcome in Children With Single Ventricle Physiology
Brief Title: Single Ventricle Outcome
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Robert Campbell, MD, Principal Investigator, Emory University
Other Study IDs: 0604-2005
Record Dates: First submitted 2006-03-27; First posted 2006-03-29 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Heart Disease, Congenital; Single Ventricle; Hypoplastic Left Heart Syndrome
Keywords: Heart Disease, Congenital; Single Ventricle; Hypoplastic Left Heart Syndrome
MeSH Terms: conditions — Heart Defects, Congenital; Univentricular Heart; Hypoplastic Left Heart Syndrome

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The objective of this research proposal is to perform an ongoing single institution prospective clinical trial examining the overall clinical outcome of children with single ventricle physiology.

DETAILED DESCRIPTION:
Congenital disease is the most common cause for infant death from a birth defect. Approximately 30,000 infants are born each year with congenital heart defects.Over one-third of those babies will require cardiac surgery. A particularly lethal cardiac defect is one with single ventricle physiology. The objective of this research proposal is to perform an ongoing single institution prospective clinical trial examining the overall clinical outcome of children with single ventricle physiology.

ELIGIBILITY:
Inclusion Criteria:

* All patients with single ventricle physiology scheduled for ultimate Fontan surgical palliation at Children's Healthcare of Atlanta will be eligible.
* All subjects must sign informed consent prior to enrollment in study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2005-06; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Campbell, MD, Principal Investigator — Associate Professor, Emory University School of Medicine
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States